CLINICAL TRIAL: NCT04845204
Title: Effects of Progressive Muscle Relaxation Techniques on Pain, Sleeping Quality and Functional Levels After Total Knee Arthroplasty
Brief Title: Relaxation Treatment in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HANDE GUNEY, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 15/77-22
Record Dates: First submitted 2021-04-06; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Relaxation; Joint; Total Knee Arthroplasty; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation Treatment (Active Comparator): Relaxation treatment (RT) is applied additional to standard physiotherapy treatment. RT includes 8 sessions (2 times a day, for four days after surgery) of relaxation exercises.
  Interventions: Other: Standard Exercises
- Standard Exercises (Active Comparator): Standard postoperative rehabilitation program is applied to Control Group. Knee-based exercises were undertaken in supine (active- assisted knee flexion using a bandage, inner range quadriceps contractions, and straight-leg raises), seated (active-assisted knee flexion using the contralateral limb and inner range quadriceps contractions), and standing (hip and knee flexion, active hamstring curls, lunges on a step, hamstring stretches) postures.
  Interventions: Other: Relaxation Treatment

INTERVENTIONS:
Other: Relaxation Treatment — Relaxation Group recieve progressive muscle relaxation exercises additional to the standard exercises. The relaxation exercises are applied two times a day till the discharge day starting on the postoperative day one. Progressive muscle relaxation included the relaxing of different muscle groups along with deep breathing. The maximal contraction period consist of the contraction of muscle groups around ankle, calf, knee, hip, lumbar, thoracic and cervical regions, shoulder, arm, forearm for 5 s and continued with a relaxation period for 30 s while focusing on breathing. These two periods ware repeated for each muscle groups and lasted approximately 30 min
  Other Names: Standard Exercises
  Arms: Standard Exercises
Other: Standard Exercises — The physiotherapy protocol is applied under the supervision of the same physiotherapist within a progressive manner immediately after surgery. Continued passive range of motion is applied twice a day starting with 45º of knee flexion range of motion and increased gradually as tolerated. All patients performed same isometric, isotonic and active exercises. Patients were instructed to bear weight as tolerated on the postoperative day 1
  Other Names: Relaxation Treatment
  Arms: Relaxation Treatment

SUMMARY:
Surgical techniques and treatment methods of the arthroplasty have been improved and the results after total knee arthroplasty (TKA) are generally good. However, some patients have suboptimal postoperative results with respect to pain and physical functioning and may not be satisfied with the results of their TKA. Psychological symptoms were found to be associated with these suboptimal results. The aim of the present study is to determine weather relaxation techniques had beneficial effects on pain, sleeping quality, functional status and physiological symptoms in TKA patients during their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis, Female Patients who are scheduled for unilateral Total Knee Arthroplasty surgery, were included in the study.

Exclusion Criteria:

* having a previous knee or hip surgery or fracture, diagnosis of rheumatoid arthritis, severe obesity (BMI>40 kg/m2), sensory and motor disorders in the operated limb, inability to understand pain assessment.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Pain Level Change | Mean change from Postoperative day 1 to day 4 recorded
  Visual analog scale

SECONDARY OUTCOMES:
Sleep Quality Change | Mean change from Postoperative day 1 to day 4 recorded
  Visual analog scale
Functional Outcomes Change | Mean change from Postoperative day4 to 6 weeks following surgery recorded
  Timed Up and Go
Functional Outcomes Change | Mean change from Postoperative day4 to 6 weeks following surgery recorded
  Western Ontario McMaster Universities Osteoarthritis Index (WOMAC)
Knee Range of Motion Change | Mean change from Postoperative day4 to 6 weeks following surgery recorded
  Flexion and Extension

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koken M, Guclu B. The Effects of Total Knee Arthroplasty on Sleep Quality. Malays Orthop J. 2019 Jul;13(2):11-14. doi: 10.5704/MOJ.1907.002. PMID 31467645
- [Background] Schache MB, McClelland JA, Webster KE. Does the addition of hip strengthening exercises improve outcomes following total knee arthroplasty? A study protocol for a randomized trial. BMC Musculoskelet Disord. 2016 Jun 13;17:259. doi: 10.1186/s12891-016-1104-x. PMID 27295978